CLINICAL TRIAL: NCT06668805
Title: A Phase 2, Randomized, Human Growth Hormone-Controlled, Multicenter, Basket Study of Vosoritide in Children With Turner Syndrome, Short Stature Homeobox-Containing Gene Deficiency, and Noonan Syndrome With an Inadequate Response to Human Growth Hormone. (CANOPY NS, TS, SHOX-D-2)
Brief Title: A Phase 2 Basket Study of Vosoritide in Children With Turner Syndrome, SHOX Deficiency and Noonan Syndrome With an Inadequate Response to Human Growth Hormone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111-211
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Short Stature Homeobox- Containing Gene SHOX Deficiency; Noonan Syndrome; Turner Syndrome
Keywords: Short Stature; Musculoskeletal Diseases; Bone Diseases; Developmental Endocrine System Diseases Natriuretic Peptide, C-Type
MeSH Terms: conditions — Noonan Syndrome; Turner Syndrome; Dwarfism; Musculoskeletal Diseases; Bone Diseases | interventions — vosoritide; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vosoritide Dose 1 - Low Dose (Experimental): Drug: Vosoritide - Dose 1 Injection
  • Experimental Drug Lyophilized powder for reconstitution
  Interventions: Drug: Vosoritide Injection
- Vosoritide Dose 2 - Medium Dose (Experimental): Drug: Vosoritide - Dose 2 Injection
  • Experimental Drug Lyophilized powder for reconstitution
  Interventions: Drug: Vosoritide Injection
- Vosoritide Dose 3- High Dose (Experimental): Drug: Vosoritide Dose 3 Injection
  • Experimental Drug Lyophilized powder for reconstitution
  Interventions: Drug: Vosoritide Injection
- Human Growth Hormone (Active Comparator): Drug: Human Growth Hormone
  Interventions: Drug: Human Growth Hormone

INTERVENTIONS:
Drug: Vosoritide Injection — Modified recombinant human C-type natriuretic peptide Vosoritide
  Arms: Vosoritide Dose 1 - Low Dose; Vosoritide Dose 2 - Medium Dose; Vosoritide Dose 3- High Dose
Drug: Human Growth Hormone — Commercial product containing somatotropin.
  Arms: Human Growth Hormone

SUMMARY:
The purpose of this basket study in children with Turner syndrome, SHOX deficiency, and Noonan syndrome is to evaluate the effect of 3 doses of vosoritide versus hGH on growth as measured by AGV after 6 months of treatment. The long-term efficacy and safety of vosoritide at the therapeutic dose will be evaluated up to FAH.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, active-controlled, multicenter, basket study of vosoritide in children with Turner syndrome, short stature homeobox-containing gene (SHOX) deficiency, or Noonan syndrome who have an inadequate response to human growth hormone (hGH) treatment. The study is intended to characterize the short-term efficacy and safety of 3 dosing regimens of vosoritide versus hGH. The efficacy and safety of the vosoritide therapeutic dose will be further evaluated, with a comparison to hGH after 2 years of treatment, and an analysis of the impact of vosoritide on final adult height (FAH).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 3 years old, and < 11 years old (females) or < 12 years old (males), at the time of signing the informed consent form
2. A genetically confirmed diagnosis of Turner syndrome, SHOX deficiency or Noonan syndrome.
3. A height assessment corresponding to a height Z-score of > -2.00 SDs and ≤ -1.75 SDs (up to 20% of participants)/≤ -2.00 SDs (at least 80% of participants) in reference to the general population of the same age and sex.
4. Tanner Stage 1, at time of signing the ICF.
5. Have been receiving continuous hGH for the treatment of short stature associated with their condition for a minimum of 1 year immediately prior to enrollment and be receiving a dose of ≥ 0.35 mg/kg weekly, with no weight-based dosing changes in the last 6 months and none planned in the future.
6. Are willing to continue on hGH at their current dose for the Baseline Growth Phase, and for 2 years post randomization if randomized to the hGH arm.
7. Inadequate response to prior hGH treatment.

Exclusion Criteria:

1. Participants with Turner syndrome known to have Y-chromosome material unless they have undergone gonadectomy and have fully external female genitalia.
2. Diagnosis of systemic disease or condition that may cause short stature other than Turner syndrome, SHOX deficiency, or Noonan syndrome, eg, renal, neoplastic, pulmonary, cardiac, gastrointestinal, immunologic and metabolic disease.
3. Bone age advanced beyond chronological age by more than 2 years.
4. Uncorrected congenital heart disease which places the participant at increased risk of an adverse cardiac outcome in the setting of hypotension,
5. Have an unstable condition likely to require surgical intervention during the study.
6. Evidence of decreased growth velocity (AGV < 1.5 cm/year) as assessed over a period of at least 6 months and growth plate closure assessed using bilateral lower extremity X-rays.
7. Previous limb-lengthening surgery, or planned or expected to have limb lengthening surgery during the study period.
8. Planned or expected bone-related surgery (ie, surgery involving disruption of bone cortex, excluding tooth extraction), during the study period.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participants must be ≥ 3 years old, and <11 years old (female) or <12 years old (males) at the time of signing the informed consent form (ICF).
Enrollment: 72 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2041-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Annualized Growth Velocity (AGV) | At 6 months

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Until the end of the study, up to 15 years
Incidence of new diagnosis of hypertrophic cardiomyopathy in children with Noonan syndrome | Every 12 months through the end of the study, up to 15 years
Incidence of cardiac conditions requiring discontinuation of study treatment | Every 12 months through the end of the study, up to 15 years
Change from baseline in height | At 6 months and at 24 months
Change from baseline in height Z-score | At 6 months and at 24 months
Change from baseline in 12-month interval AGV | 24 months
Change from baseline in upper to lower body segment ratio | At 12 and 24 months
Change from baseline in arm span to height ratio | At 12 and 24 months
Change from baseline in height up to Final Adult Height (FAH) | Every 6 months through the end of the study, up to 15 years
Change from baseline in height Z-score up to FAH | Every 6 months through the end of the study, up to 15 years
12-month interval AGV summarized by age and sex up to FAH | Every 12 months through the end of the study, up to 15 years
Tanner stage over the course of the study | Every 6 months through the end of the study, up to 15 years
Time vosoritide is present at maximum concentration (Tmax) | Every 6 months through the end of the study, up to 15 years
Maximum vosoritide observed plasma concentration (Cmax) | Every 6 months through he end of the study, up to15 years
Area under the plasma vosoritide concentration time-curve from time 0 to the last measurable concentration (AUC0-t) | Every 6 months through the end of the study, up to 15 years
Area under the plasma vosoritide concentration time-curve from time 0 to infinity (AUC0-∞) | Every 6 months through the end of the study, up to 15 years
Elimination half-life of vosoritide (t½) | Every 6 months through the end of the study, up to 15 years
Apparent clearance of vosoritide (CL/F) | Every 6 months through the end of the study, up to 15 years
Apparent volume of distribution of vosoritide (Vz/F) | Every 6 months through the end of the study, up to 15 years
Change from pre-dose in urine cyclic guanine monophosphate (cGMP) | Every 6 months through the end of the study, up to 15 years
Change from baseline in serum collagen X marker (CXM) | Every 6 months through the end of the study, up to 15 years
Change from baseline in bone age/chronological age | Every 12 months through the end of the study, up to 15 years
Change from baseline in total body (less head) BMD Z-score | Every 12 months through the end of the study, up to 15 years
Change from baseline in lumbar spine bone mineral density (BMD) Z-score | Every 12 months through the end of the study, up to 15 years
Change from baseline in total body (less head) bone mineral content (BMC) | Every 12 months through the end of the study, up to 15 years
Change from baseline in lumbar spine BMC | Every 12 months through the end of the study, up to 15 years
Change in bone morphology based on whole length lower extremity X-rays | Every 6 months through the end of the study, up to 15 years
Incidence of bone-related events of special interest (fracture, slipped capital femoral epiphysis and avascular necrosis or osteonecrosis) | Throughout study
Change from baseline in the physical domain score and total score of the QoLISSY | At 24 months
Change from baseline in the physical and social domain scores and total score of the PedsQL | At 24 months
Change from baseline in PGI-S and CaGI-S item scores | At 24 months
PGI-C and CaGI-C item scores | At 24 months
Change from baseline in PROMIS-SF Physical Activity score | At 24 months
Change from baseline in KABC-II NVI scores | At 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, PhD, Study Director — BioMarin Pharmaceutical
Locations (20):
- United States (13):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Delaware (Alfred I. Dupont Hospital for Children), Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - St. Luke's Children's Endocrinology and Diabetes, Boise, Idaho
  - Kentucky Children's Hospital, Lexington, Kentucky
  - New York Medical College, Boston, Massachusetts
  - M Health Fairview Pediatric Specialty Clinic - Explorer, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston (UT Health), Houston, Texas
- France (5):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Angers University Hospital Center, Angers, Maine-et-Loire
  - CHU de Toulouse - Hôpital des Enfants, Toulouse, Occitanie
  - South Paris University Hospitals - Bicetre Hospital, Le Kremlin-Bicêtre, Paris
  - Hôpital Robert-Debré, Paris, Paris
- IRCCS Istituto Giannina Gaslini, Genova, Genoa, Italy
- Central University Hospital of Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No